CLINICAL TRIAL: NCT00396565
Title: A Placebo-Controlled Double Blind Comparative Study of JNS007ER in Patients With Schizophrenia
Brief Title: A Study to Evaluate Effectiveness and Safety of ER OROS Paliperidone in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR012625; JNS007ER-JPN-S31 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2006-11-03; First posted 2006-11-07 (Estimated); Results first posted 2012-07-03 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; JNS007ER; Positive and Negative Syndrome Scale (PANSS); Paliperidone; Extended Release Osmotic Controlled-Release Oral Delivery System (OROS) paliperidone
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- ER OROS paliperidone (Experimental): Extended Release (ER) Osmotic Controlled-Release Oral Delivery System (OROS) paliperidone
  Interventions: Drug: ER OROS paliperidone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Olanzapine (Active Comparator)
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: ER OROS paliperidone — Type= exact number, unit= mg, number= 3, form= tablet, route= oral use. Two tablets once daily for 6 weeks.
  Arms: ER OROS paliperidone
Drug: Placebo — Form= tablet, route= oral use. Two tablets once daily for 6 weeks.
  Arms: Placebo
Drug: Olanzapine — Type= exact number, unit= mg, number= 2.5, form= tablet, route= oral use. Four tablets once daily for 6 weeks.
  Arms: Olanzapine

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of Extended Release Osmotic Controlled-Release Oral Delivery System (OROS) Paliperidone compared to placebo in patients with Schizophrenia. Olanzapine will be used as a reference drug in the study.

DETAILED DESCRIPTION:
This is a multicenter, double blind (neither the patient nor the physician knows whether drug or placebo is being taken, or at what dosage), randomized (patients are assigned different treatments based on chance), placebo- and active-controlled, parallel-group study. Patients will be randomized into 1 of 3 treatment groups to receive oral dosages of Extended Release (ER) Osmotic Controlled-Release Oral Delivery System (OROS) paliperidone 6 mg, olanzapine 10 mg, or placebo. They will receive two capsules of Paliperidone ER 3 mg, placebo or Olanzapine 5 mg once daily after breakfast for 6 weeks. The study will include a screening period, followed by double-blind treatment for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given their own consent in writing to participate in the study
* Patients diagnosed with schizophrenia according to the diagnostic criteria of DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, 295.30, 295.10, 295.20, 295.90, 295.60)
* Patients who have acute symptoms of schizophrenia
* Both inpatients and outpatients are acceptable

Exclusion Criteria:

* A DSM-IV (Diagnostic and Statistical Manual of Mental Disorders) of a mental disease diagnosis other than schizophrenia
* A DSM-IV diagnosis of substance-related disorder (except nicotine dependence and caffeine dependence) within 180 days before the screening test
* Total PANSS (Positive and Negative Syndrome System) score at the screening test <70 or >120
* Patients treated with three or more types of antipsychotic within 28 days before the screening test
* Parkinson's disease (except for those with drug-induced extra pyramidal symptoms)
* Patients with a complication of or a past history of cerebrovascular accident
* Patients with a complication of or a past history of diabetes mellitus

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2006-07; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (56):
- Japan (56):
  - Aizu-Wakamatsu
  - Fujioka
  - Fujisawa
  - Fukui
  - Hadano
  - Himeji
  - Hiratsuka
  - Hiroshima
  - Ibaraki
  - Ichikawa
  - Iida
  - Inazawa
  - Itoman
  - Kaizuka
  - Kanzaki
  - Kashihara
  - Kitakyushu
  - Kochi
  - Kōshi
  - Kumamoto
  - Kurayoshi
  - Matsudo
  - Matsusaka
  - Moriguchi
  - Morioka
  - Nagoya
  - Naha
  - Nakagami
  - Nankoku
  - Nishinomiya
  - Noda
  - Numazu
  - Ohta
  - Okinawa
  - Oyama
  - Ōita
  - Sakai
  - Sapporo
  - Takasaki
  - Takatsuki
  - Tanba
  - Tokyo
  - Tottori
  - Toyama
  - Toyoake
  - Toyonaka
  - Tōgane
  - Tsuyama
  - Ueda
  - Urasoe
  - Uruma
  - Yanagawa
  - Yao
  - Yokkaichi
  - Yokohama
  - Yokosuka

REFERENCES:
- See also: A Study to Evaluate Efficacy and Safety of ER OROS Paliperidone in Patients With Schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=412&filename=CR012625_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Informed Consent was obtained from 394 patients. The actual number of patients randomized in the study was 321. 2 subjects discontinued before treatment. 319 subjects were treated and analyzed for safety. 318 subjects were analyzed for baseline characteristics and efficacy.
Groups:
- Paliperidone Extended Release (ER) (JNS007ER): Two paliperidone ER (JNS007ER) 3 mg tablets once daily for 6 weeks
- Placebo: Two placebo tablets once daily for 6 weeks
- Olanzapine: Four olanzapine 2.5 mg tablets once daily for 6 weeks
Period: Overall Study
Arm/Group | Paliperidone Extended Release (ER) (JNS007ER) | Placebo | Olanzapine
Started | 136 | 138 | 47
Completed | 88 | 47 | 30
Not Completed | 48 | 91 | 17
Not completed — Physician Decision | 3 | 1 | 2
Not completed — Adverse Event | 5 | 13 | 3
Not completed — Withdrawal by Subject | 8 | 13 | 1
Not completed — Lack of Efficacy | 32 | 64 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paliperidone Extended Release (ER) (JNS007ER) | Placebo | Olanzapine | Total
Number analyzed (Participants) | 134 | 138 | 46 | 318
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (14.7) | 46.2 (15.1) | 46.2 (13.2) | 45.3 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 66 | 27 | 157
  Male | 70 | 72 | 19 | 161
Total Positive and Negative Syndrome Scale (PANSS) score [Mean (Standard Deviation); unit: scores on a scale] — PANSS is a medical scale that assesses various symptoms of schizophrenia. Symptoms are rated on a 7-point scale from 1 (absent) to 7 (extreme psychopathology). Total score is the sum of all 30 PANSS items, with a range of 30 (absent) to 210 (extreme ill).
  scores on a scale | 92.0 (12.9) | 91.0 (11.2) | 94.1 (12.6) | 91.9 (12.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Total Positive and Negative Syndrome Scale (PANSS).
Description: PANSS is a medical scale that assesses various symptoms of schizophrenia. The symptoms are rated on a 7-point scale from 1 (absent) to 7 (extreme psychopathology). The total score is the sum of all 30 PANSS items, with a range of 30 (absent) to 210 (extreme ill).
Time Frame: Baseline and 6 weeks
Population: Full Analysis Set excludes subjects who didn't receive test drug or didn't have post-treatment efficacy data. The Olanzapine (OLZ) group was set as an active drug group to examine clinical position of paliperidone (PAL) ER, and the superiority or non-inferiority of PAL ER 6mg to OLZ 10mg wasn't verified. LOCF imputation method was applied.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Paliperidone Extended Release (ER) (JNS007ER) | Placebo | Olanzapine
Number analyzed (Participants) | 134 | 138 | 46
scores on a scale | -9.1 (18.39) | 3.8 (18.88) | -9.9 (16.83)
Statistical Analysis 1: Comparison: Paliperidone Extended Release (ER) (JNS007ER) vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with treatment as a factor and baseline score as a covariate; Least squares mean difference = -12.7, 95% CI [-17.16 to -8.25], Standard Error of Mean 2.26

2. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) - Positive Subscale Score
Description: The PANSS Positive Subscale assesses seven positive-symptoms of schizophrenia. Positive symptoms refer to an excess or distortion of normal functions. The symptoms are rated on a 7-point scale, with a range of 7 (absent) to 49 (extreme psychopathology).
Time Frame: Baseline and 6 weeks
Population: Full Analysis Set excludes subjects who didn't receive test drug or didn't have post-treatment efficacy data. The Olanzapine(OLZ) group was set as an active drug group to examine clinical position of paliperidone(PAL) ER, and the superiority or non-inferiority of PAL ER 6mg to OLZ 10mg wasn't verified. LOCF imputation method was applied.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Paliperidone Extended Release (ER) (JNS007ER) | Placebo | Olanzapine
Number analyzed (Participants) | 134 | 138 | 46
scores on a scale | -2.6 (5.69) | 1.6 (5.53) | -2.4 (5.34)
Statistical Analysis 1: Comparison: Paliperidone Extended Release (ER) (JNS007ER) vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with treatment as a factor and with baseline score as a covariate; Least squares mean difference = -3.8, 95% CI [-5.17 to -2.51], Standard Error of Mean 0.68

3. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) - Negative Subscale Score
Description: The PANSS Negative Subscale assesses seven negative-symptoms of schizophrenia. Negative symptoms represent a diminution or loss of normal functions. The symptoms are rated on a 7-point scale, with a range of 7 (absent) to 49 (extreme psychopathology).
Time Frame: Baseline and 6 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Paliperidone Extended Release (ER) (JNS007ER) | Placebo | Olanzapine
Number analyzed (Participants) | 134 | 138 | 46
scores on a scale | -2.4 (5.05) | 0.0 (5.02) | -2.8 (4.27)
Statistical Analysis 1: Comparison: Paliperidone Extended Release (ER) (JNS007ER) vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with treatment as a factor and with baseline score as a covariate; Least squares mean difference = -2.5, 95% CI [-3.71 to -1.33], Standard Error of Mean 0.60

4. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) - General Psychopathology Subscale Score
Description: The PANSS General Psychopathology Subscale Score assesses 16 general psychopathology symptoms. The symptoms are rated on a 7-point scale, with a range of 16 (absent) to 112 (extreme psychopathology).
Time Frame: Baseline and 6 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Paliperidone Extended Release (ER) (JNS007ER) | Placebo | Olanzapine
Number analyzed (Participants) | 134 | 138 | 46
scores on a scale | -4.1 (9.52) | 2.2 (10.71) | -4.7 (9.00)
Statistical Analysis 1: Comparison: Paliperidone Extended Release (ER) (JNS007ER) vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with treatment as a factor, and with baseline score as a covariate; Least squares mean difference = -6.2, 95% CI [-8.58 to -3.80], Standard Error of Mean 1.21

5. Secondary Outcome: Proportion of Responders (≥30% Decrease in Total Positive and Negative Syndrome Scale [PANSS])
Description: Responders are subjects with 30% or more reduction from baseline in total PANSS score. PANSS is a medical scale that assesses various symptoms of schizophrenia. The symptoms are rated on a 7-point scale from 1 (absent) to 7 (extreme psychopathology). The total score is the sum of all 30 PANSS items, with a range of 30 (absent) to 210 (extreme ill).
Time Frame: Baseline and 6 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Paliperidone Extended Release (ER) (JNS007ER) | Placebo | Olanzapine
Number analyzed (Participants) | 134 | 138 | 46
Percentage of participants | 25.4 | 9.4 | 26.1
Statistical Analysis 1: Comparison: Paliperidone Extended Release (ER) (JNS007ER) vs Placebo; Test type: Superiority or Other; p = 0.0007, Fisher Exact

6. Secondary Outcome: Change From Baseline in Clinical Global Impression Scale (CGI-S)
Description: The CGI-S rating scale is a 7-point global assessment with scores as follows: 1 - Not ill, 2 - Very Mild, 3 - Mild, 4 - Moderate, 5 - Marked, 6 - Severe, and 7 - Extremely Severe.
Time Frame: Baseline and 6 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Paliperidone Extended Release (ER) (JNS007ER) | Placebo | Olanzapine
Number analyzed (Participants) | 134 | 138 | 46
scores on a scale | -0.4 (0.09) | 0.2 (0.09) | -0.3 (0.14)
Statistical Analysis 1: Comparison: Paliperidone Extended Release (ER) (JNS007ER) vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with treatment as a factor, and baseline score as a covariate; Least squares mean difference = -0.6, 95% CI [-0.84 to -0.34], Standard Error of Mean 0.13

ADVERSE EVENTS:
Arm/Group | Paliperidone Extended Release (ER) (JNS007ER) | Placebo | Olanzapine
Serious Adverse Events (participants affected / at risk) | 4/134 | 1/138 | 2/47
Other Adverse Events (participants affected / at risk) | 109/134 | 110/138 | 40/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Extended Release (ER) (JNS007ER) (N=134) | Placebo (N=138) | Olanzapine (N=47)
schizophrenia (Psychiatric disorders) | 3 | 1 | 1
pneumonia (Infections and infestations) | 1 | 0 | 0
mood altered (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Extended Release (ER) (JNS007ER) (N=134) | Placebo (N=138) | Olanzapine (N=47)
schizophrenia (Psychiatric disorders) | 22 | 59 | 11
Insomnia (Psychiatric disorders) | 15 | 14 | 5
Nasopharyngitis (Infections and infestations) | 14 | 11 | 1
Blood creatine phosphokinase increased (Investigations) | 9 | 8 | 2
Constipation (Gastrointestinal disorders) | 11 | 2 | 5
Weight increased (Investigations) | 8 | 0 | 5
Blood triglycerides increased (Investigations) | 9 | 0 | 3
Extrapyramidal disorder (Nervous system disorders) | 10 | 1 | 1
Somnolence (Nervous system disorders) | 3 | 1 | 8
Pyrexia (General disorders) | 5 | 3 | 3
Basophil count increased (Investigations) | 1 | 8 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 7 | 1 | 1
Thirst (General disorders) | 2 | 2 | 5
Dizziness (Nervous system disorders) | 1 | 2 | 3
White blood cell count increased (Investigations) | 2 | 1 | 3
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 3
Tachycardia (Cardiac disorders) | 1 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Without prior notification to the sponsor, the PI cannnot dislose trial results and related documents of trials to a third party.